CLINICAL TRIAL: NCT03353194
Title: The Canadian Cerebral Palsy Registry - Le Registre Canadien de la Paralysie Cérébrale
Brief Title: Canadian CP Registry - Registre Canadien de la Paralysie Cérébrale
Status: Completed | Type: Observational
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: Kids Brain Health Network (Unknown); Children's Treatment Network (Network); Montreal Children's Hospital of the MUHC (Other); Alberta Children's Hospital (Other); Women and Children's Health Research Institute, Canada (Other); Provincial Health Services Authority British Columbia (Other); IWK Health Centre (Other); The Hospital for Sick Children (Other); Holland Bloorview Kids Rehabilitation Hospital (Other)
Responsible Party: Principal Investigator, Maryam Oskoui, MD, MSc, FRCPC, FAAN, Associate Professor, Departments of Pediatrics and Neurology & Neurosurgery, McGill University Health Centre/Research Institute of the McGill University Health Centre
Other Study IDs: 09-234-PED
Record Dates: First submitted 2017-11-15; First posted 2017-11-27 (Actual); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: Cerebral Palsy
Keywords: Cerebral Palsy; Canada; Registry
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Canadian Cerebral Palsy (CP) Registry is a confidential, nation-wide collection of medical and social information about children with cerebral palsy. The Registry was first implemented in 2003 in 6 administrative regions of Quebec and was later extended to paediatric centres in Newfoundland, Nova Scotia, Ontario, Alberta, and British Columbia. Over 1850 children living with Cerebral Palsy have been registered so far. The Registry is the first national registry for cerebral palsy in North America.

DETAILED DESCRIPTION:
The Canadian Cerebral Palsy Registry is a multi-regional Canadian registry to identify potential risk factors related to pregnancy and interactions of the environment and genetics. The Registry provides researchers with the approximate number of children with cerebral palsy across Canada, and data in the Registry helps researchers explore reasons behind the causes of cerebral palsy, in addition to supporting studies which may lead to improvements in the overall care of children with CP.

Cerebral palsy is the most common cause of physical disability in children in Canada and it is important that we gain a better understanding of its prevalence, risk factors and current clinical profile. The Canadian CP Registry provides valuable data from different Canadian regions which can be shared and analyzed so as to provide answers to these important questions. Specifically, the Registry serves to:

* Characterize the profile of children living with CP across the country
* Identify risk factors associated with CP
* Monitor the prevalence of CP across the country
* Provide a platform for subject recruitment for population-based research on CP

ELIGIBILITY:
Inclusion Criteria:

* Under 18 (age cut-off varies by region)
* Diagnosed with Cerebral Palsy
* Living in Canada

Exclusion Criteria:

* Uncertain CP diagnosis

Ages: 18 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children living with a diagnosis of Cerebral Palsy in Canada.
Sampling Method: Probability Sample
Enrollment: 2771 (Actual)
Dates: Start 2004-04-14 (Actual); Primary Completion 2020-04 (Actual); Study Completion 2020-04 (Actual)

PRIMARY OUTCOMES:
Characterize the CP profile across Canada | An average of every two years, up to study completion or ten years, whichever comes first.
  CP subtype, severity, and associated conditions

CONTACTS AND LOCATIONS:
Overall Officials: Michael I Shevell, MDCM, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre; Maryam Oskoui, MD, MSc, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (15):
- Canada (15):
  - Alberta Children's Hospital, Calgary, Alberta
  - Glenrose Rehabilitation Hospital, Edmonton, Alberta
  - Sunny Hill Health Centre for Children, Vancouver, British Columbia
  - Janeway Health Center, St. John's, Newfoundland and Labrador
  - IWK Health Centre, Halifax, Nova Scotia
  - Children's Treatment Network, Barrie, Ontario
  - Holland-Bloorview Kids Rehabilitation Hospital, Toronto, Ontario
  - Centre régional de réadaptation La RessourSe, Gatineau, Quebec
  - Centre de réadaptation Le Bouclier, Joliette, Quebec
  - Centre de Réadaptation Marie-Enfant, Montreal, Quebec
  - MAB-Mackay Rehabilitation Centre, Montreal, Quebec
  - Montreal Children's Hospital, Montreal, Quebec
  - Shriners Hospital Montreal, Montreal, Quebec
  - Institut de réadaptation physique du Québec, Québec, Quebec
  - Centre de réadaptation Estrie, Sherbrooke, Quebec

REFERENCES:
- [Result] Oskoui M, Gazzellone MJ, Thiruvahindrapuram B, Zarrei M, Andersen J, Wei J, Wang Z, Wintle RF, Marshall CR, Cohn RD, Weksberg R, Stavropoulos DJ, Fehlings D, Shevell MI, Scherer SW. Clinically relevant copy number variations detected in cerebral palsy. Nat Commun. 2015 Aug 3;6:7949. doi: 10.1038/ncomms8949. PMID 26236009
- [Result] Oskoui M, Messerlian C, Blair A, Gamache P, Shevell M. Variation in cerebral palsy profile by socio-economic status. Dev Med Child Neurol. 2016 Feb;58(2):160-6. doi: 10.1111/dmcn.12808. Epub 2015 May 22. PMID 26010819
- [Result] Shevell M, Dagenais L, Oskoui M. The epidemiology of cerebral palsy: new perspectives from a Canadian registry. Semin Pediatr Neurol. 2013 Jun;20(2):60-4. doi: 10.1016/j.spen.2013.06.008. No abstract available. PMID 23948680
- [Result] Oskoui M, Majnemer A, Dagenais L, Shevell MI. The relationship between gross motor function and manual ability in cerebral palsy. J Child Neurol. 2013 Dec;28(12):1646-52. doi: 10.1177/0883073812463608. Epub 2012 Oct 30. PMID 23112248
- [Result] Garfinkle J, Wintermark P, Shevell MI, Oskoui M. Children born at 32 to 35 weeks with birth asphyxia and later cerebral palsy are different from those born after 35 weeks. J Perinatol. 2017 Aug;37(8):963-968. doi: 10.1038/jp.2017.23. Epub 2017 Mar 16. PMID 28300820
- [Result] Oskoui M, Joseph L, Dagenais L, Shevell M. Prevalence of cerebral palsy in Quebec: alternative approaches. Neuroepidemiology. 2013;40(4):264-8. doi: 10.1159/000345120. Epub 2013 Jan 24. PMID 23363886